CLINICAL TRIAL: NCT05436457
Title: Multi-site External Validation and Improvement of a Clinical Screening Tool for Future Firearm Violence
Brief Title: Clinical Screening for Firearm Violence Risk
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jason E. Goldstick, Research Associate Professor, University of Michigan
Other Study IDs: HUM00188023; 1R01CE003294-01 (NIH)
Record Dates: First submitted 2022-06-22; First posted 2022-06-29 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Firearm Injury
Keywords: Injury Prevention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 18-24 Year Olds in Emergency Department: Individuals age 18-24 recruited from one of the four study sites in Flint (1 hospital), Seattle (1 hospital), and Philadelphia (2 hospitals)

SUMMARY:
The purpose of the proposed work is to harness cutting-edge machine learning methods to optimize prediction of future firearm violence in youth ages 18-24 so that prevention resources can be allocated efficiently.

DETAILED DESCRIPTION:
Firearm violence is a public health crisis in the United States, and new epidemiological data suggest we may have reached a new endemic level of firearm mortality in recent years. Youth are disproportionately affected by firearm violence, with those age 18-24 being demonstrably the highest risk group. This study will recruit 1,500 youth age 18-24 from urban emergency departments (EDs) in three broadly different locales-Flint, Philadelphia, and Seattle-and administer a baseline survey covering several domains of potential risk factors for future violence, and follow up with those youth at 6- and 12-months to ascertain the primary outcome-firearm violence involvement (as victim or perpetrator, including threats and sub-clinical injuries)-as well as the secondary outcomes: high-risk firearm behaviors, non-firearm violence, and violent injury. This work will generate new insights into the prediction of firearm violence, and will lay the ground for future research involving the development and testing of interventions for interpersonal firearm violence both by identifying potential high-leverage modifiable predictive factors, and by focusing on youth most in need of intervention.

ELIGIBILITY:
Inclusion Criteria:

* Flint, Philadelphia, or Seattle Youth between the ages of 18-24 seeking care for any reason at Hurley Medical Center, the Hospital of University of Pennsylvania, Penn Presbyterian Medical Center, or Harborview Medical Center Emergency Department
* Can provide consent for the study

Exclusion Criteria:

* Do not understand English (<1% in prior work)
* Unable to provide consent due to mental status (e.g., alcohol intoxication, acute psychosis) or medical instability.
* ED visit requiring intensive psychosocial services (e.g., sexual assault, psychosis, active suicidal ideation, or child abuse)
* In active police custody/prisoners (as they cannot provide consent)

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Youth aged 18-24 seeking care at the Emergency departments of Hurley Medical Center, the Hospital of University of Pennsylvania, Penn Presbyterian Medical Center, or Harborview Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 1506 (Actual)
Dates: Start 2021-07-26 (Actual); Primary Completion 2024-08-22 (Actual); Study Completion 2024-08-22 (Actual)

PRIMARY OUTCOMES:
Firearm Violence Involvement | 1 Year After Baseline ED Visit
  The primary outcome for this study is firearm violence involvement, as perpetrator or victim. This will be measured in part by the Conflict Tactics Scale 2, as established by Straus et al. CTS-2 is comprised of a 6-point scale, measuring how often the respondent has experienced each type of violence, ranging from never to more than 20 times. The primary outcome here will be a binary indicator comprised of any affirmative response to the questions asked as part of items 1-3 below, or any firearm events found from the objective chart review.
  1. Two self-reported measurements of firearm violence perpetration adapted from the modified conflict tactics scale (CTS-2).
  2. Two self-reported measurements of firearm violence victimization adapted from the modified conflict tactics scale (CTS-2).
  3. Presentation to the emergency department for a firearm injury (ICD-10 codes: X72-X74, W32-W34, X93-X95), measured based on objective chart review during the one year following baseline.

SECONDARY OUTCOMES:
Risky Firearm Behaviors | 1 Year After Baseline ED Visit
  As established by Carter et al based on a) twelve items from the Tulane Youth Study that measure firearm carriage and discharge in high-risky situations (e.g., discharging a firearm while committing a crime, or carrying a firearm while using drugs); b) the four firearm violence perpetration/victimization outcomes listed under the primary outcome; and c) firearm violence threats (as victim or perpetrator), as measured by the modified conflict tactics scale (CTS-2)
Non-Firearm Violence | 1 Year After Baseline ED Visit
  22 self-reported measurements for non-firearm violence perpetration (11 for partner, 11 for non-partner) adapted from the CTS-2, 22 self-reported measurements for non-firearm violence victimization (11 for partner, 11 for non-partner) adapted from the CTS-2, and 6 items about fighting, adapted from the National Longitudinal Study of Adolescent Health.
Violent Injury | 1 Year After Baseline ED Visit
  Presentation to the emergency department for any violent injury, measured based on objective chart review during the one year following baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Jason E. Goldstick, PHD, Principal Investigator — University of Michigan
Locations (4):
- United States (4):
  - Hurley Medical Center, Flint, Michigan
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Harborview Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
After study completion, de-identified data will be curated and uploaded through the Inter-University Consortium for Political and Social Research (ICPSR) run through the University of Michigan. ICPSR stores, curates, and provides access to data generated through social research studies in service to open science, which acts in service to optimized data sharing, rigorous detailing of study methods and citations for measures, and ensuring long-term preservation of the study data. Through the data curation process, data are cleaned and standardized for use, and data documentation is rigorously developed so that data sets and the associated documentation can be understood at a basic by any potential users. The uploaded data will be de-identified to ensure no linkages to individual research participants and will exclude variables that could lead to deductive disclosure of the identity of any individual subjects.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: After the study is completed, with no specified time for when sharing will end.
Access Criteria: Registration with ICPSR and agreement to follow their rules and policies